CLINICAL TRIAL: NCT02390479
Title: Gingival Crevicular Fluid Levels of Sclerostin, Osteoprotegerin (OPG) and RANKL in Health, Disease and After Treatment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Umut BALLI (Other)
Responsible Party: Sponsor-Investigator, Umut BALLI, Bulent Ecevit University, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2013-112-01/10
Record Dates: First submitted 2015-02-18; First posted 2015-03-17 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-03

CONDITIONS: Periodontitis
Keywords: Sclerostin; OPG; RANKL
MeSH Terms: conditions — Periodontitis; Sclerosteosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic periodontitis (Active Comparator): GCF samples were taken before and after treatment chronic periodontitis patients.
  Intervention: Non- surgical periodontal treatment (SRP and oral hygiene instructions)
  Interventions: Other: non surgical periodontal treatment
- clinically healthy periodontium (Placebo Comparator): GCF samples were taken at baseline Intervention: oral hygiene instructions
  Interventions: Other: non surgical periodontal treatment

INTERVENTIONS:
Other: non surgical periodontal treatment — 1. SRP under local anaesthesia, in a total of four clinical visits
  2. Oral hygiene instructions including the modified Bass technique, regular toothpaste, and an appropriate interdental cleaning device with dental floss and interdental brush.

SUMMARY:
The primary objective of this case-control intervention study to explore the effectiveness of non surgical periodontal therapy on the gingival crevicular fluid (GCF) levels of sclerostin in patients with chronic periodontitis (CP) so as to get a more detailed insight into its diagnostic and prognostic potential as a biomarker of periodontal disease.

DETAILED DESCRIPTION:
All individuals underwent a full-mouth periodontal examination, which included probing pocket depth (PPD), clinical attachment level (CAL), plaque index (PI), gingival index (GI), bleeding on probing (BOP). Individuals were categorized into three groups: individuals with clinically healthy periodontium (group 1), patients with chronic periodontitis (group 2), and group 3 consisted of the patients with chronic periodontitis (group 2), treated by scaling and root planning. GCF samples in grup 1 were taken at baseline. In group 2, GCF samples were taken before and after non- surgical periodontal treatment. Sclerostin, OPG and RANKL levels were determined using the enzyme-linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for the healthy group were GI = 0, PPD and CAL ≤ 3 mm, and no signs of attachment and bone loss
* Criteria for the chronic periodontitis group were clinical signs of inflammation, such as red color and swelling of the gingival margin, GI ≥ 2, PPD and CAL ≥ 5 mm with bone loss (>30% of the existing teeth)

Exclusion Criteria:

* Aggressive periodontitis, systemic diseases (i.e., diabetes mellitus, cancer, human immunodeficiency virus, bone-related diseases that compromise sclerostin, OPG or RANKL levels and collagen-metabolic diseases, or disorders), chronic high-dose steroid therapy, radiation or immunosuppressive therapy, allergy or sensitivity to any drug, pregnancy, lactation, and current smoking, smoking within the past 5 years. The individuals had no history of periodontal therapy or drug therapy (e.g. anti-inflammatory, antibiotic treatment or any other pharmacological treatment) for at least six months.

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Biochemical parameters (Sclerostin levels, RANKL/OPG ratio ) | Baseline and 6 weeks after treatment
  The changes in levels of sclerostin, OPG and RANKL 6 weeks after periodontal treatment determined by ELISA. The changes in levels of sclerostin were analyzed to determine diagnostic and prognostic potential as a biomarker of periodontal disease. The relative RANKL/OPG ratio (bone resorption marker) was also calculated to detect the relationship between sclerostin levels.

SECONDARY OUTCOMES:
Probing pocket depth | Baseline and 6 weeks after treatment
  The changes in probing pocket depth after periodontal treatment.Probing pocket depth was measured for determining severity of disease and clinic outcome.
Probing pocket depth and clinical attachment level | Baseline and 6 weeks after treatment
  The changes in clinical attachment level after periodontal treatment. Clinical attachment level was measured for determining severity of disease and clinic outcome. Also, clinical attachment level was also analyzed to detect the relationship between sclerostin, OPG and RANKL levels.
Gingival index | Baseline and 6 weeks after treatment
  The changes in gingival index after periodontal treatment. Gingival index was recorded for classifying and evaluating (coronally) gingival inflammation. Also, gingival index was also analyzed to detect the relationship between sclerostin, OPG and RANKL levels.
Plaque index | Baseline and 6 weeks after treatment
  The changes in plaque index after periodontal treatment. Plaque index was recorded for determining and classifying oral hygiene status.
Bleeding on probing | Baseline and 6 weeks after treatment
  The changes in bleeding on probing after periodontal treatment. Bleeding on probing was recorded for classifying and evaluating (apically) gingival inflammation.